CLINICAL TRIAL: NCT05100459
Title: The Effects of Pasture-raised Versus Conventional Whey Protein Supplementation on Vascular Function and Markers of Exercise-induced Muscle Damage and Inflammation in Resistance-trained Individuals
Brief Title: The Effects of Whey Protein Supplements on Markers of Exercise-induced Muscle Damage in Resistance-trained Individuals
Acronym: WheyProtein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Mickleborough, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12559
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Muscle Damage; Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — hydroxide ion; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pasture-raised whey protein (Experimental): whey protein from strictly grass fed cows
  Interventions: Dietary Supplement: Pasture-raised whey protein
- Conventional whey protein (Experimental): whey protein from conventional animal feeding operation
  Interventions: Dietary Supplement: Conventional whey protein
- Placebo (Placebo Comparator): Maltodextrin given in iso-caloric amounts to protein
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pasture-raised whey protein — 25 grams of protein delivered 3 times daily
  Other Names: Premium Blend Protein, Pasture Raised, Grass Fed, unflavored, Muscle Feast, Nashport, OH, USA
  Arms: Pasture-raised whey protein
Dietary Supplement: Conventional whey protein — 25 grams of protein delivered 3 times daily
  Other Names: 100% Whey Protein Powder, unflavored, TGS Nutrition, Las Vegas, NV, USA
  Arms: Conventional whey protein
Dietary Supplement: Placebo — Iso-caloric placebo taken 3 times daily like the protein supplementation
  Other Names: Maltodextrin, Bulk Supplements, Henderson, NV, USA
  Arms: Placebo

SUMMARY:
Intense exercise can bring about various side effects to one's body. Less range of motion, increased pain sensitivity, increased muscle swelling, and decreased muscle strength can occur immediately after exercise. These side effects can be referred to exercise induced muscle damage (EIMD) and can sometimes last many days. This study's goal is to evaluate the effects of various protein supplements on EIMD symptoms as well as on blood vessel health during the recovery period after muscle damaging exercise.

DETAILED DESCRIPTION:
Eccentric exercise can result in exercise induced muscle damage (EIMD), which can cause an abundance of ultrastructural muscular disruption and pro-inflammatory and pro-oxidant activity in the body, leading to an impairment of muscular force production and range of motion, along with elevated pain sensitivity, increased swelling, and arterial stiffness. Pasture-raised dairy products, obtained from strictly grass-fed cows, have been shown to possess more anti-inflammatory-, antioxidant-, and antihypertensive-like biochemicals compared with conventional products (i.e., with a different nutrient composition from a diet rich in grains versus grasses). However, human research trials on these products, such as whey protein concentrate (WPC), are neglected. This study addresses this gap, with a double-blind, randomized, placebo-controlled trial that compares the effect of conventional WPC versus WPC supplementation reported to be derived from pasture-raised cows on vascular function and indirect markers of muscle damage and inflammation in response to eccentric EIMD in healthy, young, resistance-trained women and men. Thirty resistance-trained individuals will complete an intense EIMD bout consisting of eccentric barbell back squats and then will be assessed 24, 48, and 72 hours post-EIMD for muscle soreness, range of motion, maximal isometric voluntary contraction, peripheral fatigue via magnetic stimulation, countermovement jump, barbell back squat velocity, and vascular function (i.e., arterial stiffness via carotid femoral pulse wave velocity). Subjects will be grouped into a conventional WPC, pasture-raised WPC, and placebo supplementation group and consume their respective supplementation thrice daily immediately post-EIMD until the study's completion.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-40 years old
* ≥3 months uninterrupted training of ≥3 days/week of resistance training
* Self-reported to be healthy

Exclusion Criteria:

* Not within defined age range
* History of allergy to dairy products
* History of experiencing pain while exercising in the lower extremities (i.e., hips/knees)
* Current use of anti-inflammatory/anti-pain medication (i.e., nonsteroidal anti-inflammatory drugs (NSAIDs) such as Tylenol, Advil, or Aleve
* Are pregnant or could possibly be pregnant by self-report
* People who answer 'yes' to any of the pre-participation screening questions on the PAR-Q questionnaire.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Titin | Four days
  Muscle damage assessment via urinary titin via ELISA (MBS2881644, Human Titin ELISA® Kit, MyBioSource.com, Inc., San Diego, USA). Units: pmol
Isometric torque | Four days
  Isometric torque assessment of right leg extensors will be conducted at a knee angle of 90 degrees using a calibrated load cell (model Z Tension Load Cell; Dillon, Fairmont, MN) Units: Nm
Range of motion | Four days
  Hamstring flexibility and stiffness will be measured using a sit-and-reach box (Lafayette Instrument Company, Lafayette, IN) test. Units: cm
delayed onset muscle soreness | Four days
  Visual analog scale of muscle soreness (delayed onset muscle soreness; DOMS) - Knee extensor soreness will be assessed using a visual analogue scale with "no soreness" indicated at one end (score 0) and "unbearably painful" at the other (score 100). Units: arbitrary units
Pain pressure threshold | Four days
  Muscle tenderness, known as pain pressure threshold, will be quantified using a digital algometer (Force One, Wagner Instruments, Greenwich, CT) on pre-marked sites at two specific points on the quadriceps (rectus femoris-RF and vastus lateralis-VL) and one on the calf (gastrocnemius-GM). Units: percentage change from baseline
Peripheral Fatigue | Four days
  Peripheral fatigue will be assessed via magnetic stimulation (Magstim 200-2; Jali Medical, Newton, MA, USA) of the femoral nerve, which will be used to elicit a quadriceps twitch. Units: Nm
Countermovement Jump | Four days
  A linear position transducer (GymAware Powertool; Kinetic Performance Technology, Canberra, Australia) interfaced with an iPad (Apple, CA, USA) will be used to calculate countermovement jump (CMJ) height. Units: cm
Barbell back squat velocity | Four days
  The mean velocity of the barbell will be measured using the linear position transducer as per the load velocity profile relationship. Units: m/s

SECONDARY OUTCOMES:
Arterial Stiffness | Four days
  Utilizing carotid femoral pulse wave velocity via applanation tonometry, considered the non-invasive gold standard of central arterial stiffness, the ATCOR SphygmoCor® (Naperville, IL, USA) device will be utilized. Units: m/sec

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Mickleborough, Ph.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in muscle damage. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.